CLINICAL TRIAL: NCT01125176
Title: A Phase II Study of Daily Alternating Thalidomide and Lenalidomide Therapy Plus Rituximab (ThRiL) as Initial Treatment for Patients With CLL
Brief Title: Alternating Thalidomide and Lenalidomide Therapy Plus Rituximab (ThRiL) as Initial Treatment for Patients With CLL
Acronym: ThRiL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1112012062; RV-CLL-PI-0391 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2010-04-23; First posted 2010-05-18 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Thalidomide; Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): In Cycle -1, even numbered patients will receive oral lenalidomide daily on days 1-14 and then no treatment on days 15-28. In Cycle -1, odd numbered patients will receive oral thalidomide daily days 1-14 followed by no treatment on days 15-28. Starting with cycle 1, all patients will alternate daily thalidomide (every odd day) with daily lenalidomide (every even day) for days 1-28. Rituximab will be given on days 1, 8, 15, and 22 starting with Cycle 1, and then again every 6th cycle thereafter (cycles 7, 13, 19, etc.)
  Interventions: Drug: thalidomide; Drug: lenalidomide; Biological: rituximab

INTERVENTIONS:
Drug: thalidomide — 50 mg oral dosing every other day
  Other Names: Thalomid
Drug: lenalidomide — varying oral doses every other day (max 25 mg/day)
  Other Names: Revlimid
Biological: rituximab — 375 mg/m2 intravenously on days 1, 8, 15, and 22 of cycle 1. Then, repeated on days 1, 8, 15, and 22 of every 6th cycle thereafter (Cycle 7, 13, 19, etc.)
  Other Names: Rituxan

SUMMARY:
The investigators' hypothesis is that treatment of CLL with an alternating daily dosing schedule of thalidomide and lenalidomide may result in better tolerability by decreasing each agent's individual toxicities, while preserving efficacy, and therefore lead to a longer duration of therapy and improved responses. Additionally, the combination of the 2 agents may have additive or synergistic effects therapeutically.

In Cycle -1, odd numbered patients will receive oral thalidomide daily days 1-14 followed by no treatment on days 15-28. Even numbered patients will receive oral lenalidomide daily on days 1-14 and then no treatment on days 15-28. Starting with cycle 1, patients will alternate daily thalidomide (every odd day) with daily lenalidomide (every even day) for days 1-28. Rituximab will be given on days 1, 8, 15, and 22 starting with Cycle 1, and then again every 6th cycle thereafter (cycles 7, 13, 19, etc.)

DETAILED DESCRIPTION:
This is an open label, phase II, single arm, and single institution study investigating daily alternating therapy with IMiD™ compounds, thalidomide and lenalidomide, plus rituximab in untreated CLL patients requiring treatment. In order to obtain correlative samples, patients will receive a two week course of single agent thalidomide or lenalidomide before beginning treatment with the combination regimen. Half of the patients (odd numbered subjects) will start with a two week course of single agent thalidomide and the other half of the patients (even numbered subjects) will start with a two week course of single agent lenalidomide. This will allow the study of correlative samples of monotherapy with either IMiD™ agent. In Cycle -1 half of the patients (odd numbered subjects) will receive thalidomide 50mg PO daily on days 1-14, followed by no treatment days 15-28 and the other half of the patients (even numbered subjects) will receive lenalidomide PO daily on days 1-14, followed by no treatment days 15-28. Starting cycle 1: Patients will receive thalidomide 50 mg every other day (every odd day on days 1-28: Days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25 & 27 of a 28 day cycle) alternating with lenalidomide on alternate every other day, dosed based upon current level with stepwise incremental dosing (every even day on days 1-28: Days 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 & 28 of a 28 day cycle). The starting dose of lenalidomide will be based on calculated creatinine clearance and the dose of lenalidomide may be escalated as tolerated to maximal dose of 25 mg (see Section 5 for details). Rituximab 375 mg/m2 will be administered on days 1, 8, 15 and 22 starting with Cycle 1 and then again on the same weekly x 4 schedule every 6th cycle thereafter (Cycles 7, 13, 19, etc).

ELIGIBILITY:
Inclusion criteria:

1. Confirmed diagnosis of CLL or SLL based upon standard criteria as outlined in the IWCLL Update of the 1996 NCI-Working Group criteria for CLL:

a) Presence of one of the following:

1. more than or equal to 5 x 10^9 B lymphocytes/L in the peripheral blood for a duration of at least 3 months. Patients with a B lymphocytosis will be characterized as CLL, while those without will be characterized as SLL

2. the presence of lymphadenopathy resulting from infiltration with lymphocytes with the phenotype of CLL

3. bone marrow infiltration with lymphocytes with the phenotype of CLL

b) Lymphocytes with the morphologic appearance of small, mature appearing lymphocytes, with less or equal to 55 percent prolymphocytes (blood or bone marrow)

c) Cellular phenotype characterized by the:

1. co-expression of the CD5, CD20, and CD23 surface antigens
2. clonal kappa or lambda light chain expression
3. dim surface immunoglobulin expression

2. No prior therapy for CLL, including treatment for autoimmune conditions that have developed since the initial diagnosis of CLL.

3. Active disease requiring therapy as defined by the IWCLL Update of the 1996 NCIWG guidelines:

1. Evidence of progressive marrow failure as manifested by the development of worsening of anemia and / or thrombocytopenia
2. Massive, progressive, or symptomatic splenomegaly
3. Massive, progressive, or symptomatic lymphadenopathy
4. Progressive lymphocytosis with an increase of more than 50 percent over a 2-month period or a lymphocyte doubling time of less than 6 months.
5. Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroids or other standard therapy
6. Presence of disease related symptoms: unintentional weight loss of more than 10 percent within previous six months, significant fatigue, fevers greater than 100.5 F or 38.0 C for 2 or more weeks without evidence of infection, night sweats for more than 1 month without evidence of infection.

   4. Understand and voluntarily sign an informed consent form.

   5. Age at least 18 years at the time of signing the informed consent form.

   6. Able to adhere to the study visit schedule and other protocol requirements.

   7. ECOG performance status of at most 2 at study entry.

   8. Laboratory test results within these ranges:
   * Absolute neutrophil count at least 1000/mm³
   * Platelet count at least 50,000/mm³
   * Creatinine clearance of at least 30 mL/min by Cockroft-Gault formula. Patients with a baseline creatinine clearance of greater than 30 and less than 60 mL/min will have a starting dose of lenalidomide 5 mg PO every other day per the defined schedule. Patients with a baseline creatinine clearance of ≥ 60 mL/min will have a starting dose of lenalidomide 5 mg PO daily per the defined schedule.
   * Total bilirubin at most 1.5 times the ULN, unless abnormality is the result of Gilbert's disease or the result of the CLL.
   * AST (SGOT) and ALT (SGPT) at most 3 x ULN (or at most 5 x ULN if due to the CLL)

     9. Disease free of prior malignancies for at least 2 years with exception of curatively treated basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.

     10. All study participants must be registered into the mandatory Revlimid REMS and S.T.E.P.S. ( P-TAP: Protocol Therapy Assistance Program) program(s), and be willing and able to comply with the requirements of Revlimid REMS and S.T.E.P.S.

     11. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 -14 days prior to and again within 24 hours of starting treatment and again within 24 hours before the first dose of lenalidomide AND thalidomide. FCBP must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide and/or thalidomide. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS program . Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.

     12. Able to take aspirin 81 or 325 mg daily as prophylactic anticoagulation, unless already on therapeutic anticoagulation. Patients intolerant to ASA may use coumadin or low molecular weight heparin.

   Exclusion criteria:
   1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from providing informed consent.
   2. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
   3. Evidence of laboratory TLS by Cairo-Bishop Definition of Tumor Lysis Syndrome. Subjects may be enrolled upon correction of electrolyte abnormalities.
   4. Concurrent use of other anti-cancer agents or treatments.
   5. Prior treatment with thalidomide or lenalidomide.
   6. Active serious infection not controlled with antibiotics.
   7. Autoimmune hemolytic anemia or thrombocytopenia requiring treatment.
   8. Known positive for HIV
   9. Active infection with hepatitis B, defined by being positive for HepBsAg or Hep B DNA by PCR, or hepatitis C
   10. Pre-existing peripheral neuropathy greater than grade 2
   11. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide and/or thalidomide).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-03-30 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2020-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Furman, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were accrued to the study at Weill Cornell Medical College between March 2012 and September 2013.
Pre-assignment Details: One participant was deemed ineligible for the study following the completion of the informed consent process.
Groups:
- All Subjects: In Cycle -1, even numbered patients will receive oral lenalidomide daily on days 1-14 and then no treatment on days 15-28.
  In Cycle -1, odd numbered patients will receive oral thalidomide daily days 1-14 followed by no treatment on days 15-28.
  Starting with cycle 1, all patients will alternate daily thalidomide (every odd day) with daily lenalidomide (every even day) for days 1-28. Rituximab will be given on days 1, 8, 15, and 22 starting with Cycle 1, and then again every 6th cycle thereafter (cycles 7, 13, 19, etc.)
  Thalidomide: 50 mg oral dosing every other day
  Lenalidomide: varying oral doses every other day (max 25 mg/day)
  Rituximab: 375 mg/m2 intravenously on days 1, 8, 15, and 22 of cycle 1. Then, repeated on days 1, 8, 15, and 22 of every 6th cycle thereafter (Cycle 7, 13, 19, etc.)
Period: Treatment Phase
Arm/Group | All Subjects
Started | 14
Completed | 13
Not Completed | 1
Period: Post-treatment Follow-up Phase
Arm/Group | All Subjects
Started | 13
Completed | 2
Not Completed | 11

BASELINE CHARACTERISTICS:
Population: 14
Arm/Group | All Subjects
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate as Defined as the Number of Patients Who Experience a Response (Complete or Partial) to Treatment at the Time of Best Response
Description: Response will be evaluated in this study using the International Workshop on CLL (IWCLL) update of the 1996 NCI-Working Group criteria for CLL, which includes assessment of the following: clonal lymphocytes in the peripheral blood by flow cytometry, blood tests for neutrophil count, hemoglobin, and platelet count, CT examination for lymphadenopathy, hepatomegaly, splenomegaly, constitutional symptoms, bone marrow assessment via biopsy/aspirate, and evaluation for disease transformation.
Time Frame: From date of study drug initiation until date of best response, assessed up to 6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 14
Participants | 12
Statistical Analysis 1: Comparison: All Subjects; Test type: Other — Exact Clopper-Pearson 95% confidence interval for overall response rate; Proportion (percent) = 85.7, 95% CI 2-sided [73.5 to 100.0]

2. Secondary Outcome: Progression Free Survival
Description: Measured from time of study drug administration to progression or death, measured in months.
Time Frame: From date of study drug initiation until date of progression or death, whichever occurs first, assessed through study completion up to 100 months.
Population: The one not assessable came off treatment prior to having an assessment.
Measure: Median (Full Range); unit: months
Arm/Group | All Subjects
Number analyzed (Participants) | 13
months | 48 [22 to 54]

3. Secondary Outcome: Duration of Response
Description: Measured from end of treatment to progression or death, measured in months.
Time Frame: From date of end of treatment to progression or death, whichever occurs first, assessed through study completion up to 100 months.
Population: The one not assessable came off treatment prior to having an assessment.
Measure: Median (Full Range); unit: months
Arm/Group | All Subjects
Number analyzed (Participants) | 13
months | 70 [34 to 85]

4. Secondary Outcome: Time to Response
Description: Measured from time of study drug administration to initial response (partial or complete), measured in months.
Time Frame: From date of study drug initiation to date of initial response, assessed up to 12 months.
Measure: Median (Full Range); unit: months
Arm/Group | All Subjects
Number analyzed (Participants) | 14
months | 10 [3 to 12]

5. Secondary Outcome: Overall Survival
Description: Measured from time of study drug administration to death, measured in months.
Time Frame: From date of study drug initiation to date of death, assessed through study completion up to 105 months.
Measure: Median (Full Range); unit: months
Arm/Group | All Subjects
Number analyzed (Participants) | 14
months | 97 [13 to 105]

ADVERSE EVENTS:
Time Frame: From date of study drug initiation to 30 days post-date of last dose of study drug, assessed over an average of 3 years, 6 months.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 4/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=14)
Pneumonia (Infections and infestations) | 1 (14)
Acute renal insufficiency (Renal and urinary disorders) | 1 (14)
Fever (General disorders) | 1 (14)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (14)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=14)
Anemia (Blood and lymphatic system disorders) | 6
Platelet count decreased (Investigations) | 7
Lymph node pain (Blood and lymphatic system disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Blood bilirubin increased (Investigations) | 2
Lymphocyte count increased (Investigations) | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3
Fever (General disorders) | 4
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 8
Lymphocyte count decreased (Investigations) | 3
Rash (Skin and subcutaneous tissue disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Arthralgias (Musculoskeletal and connective tissue disorders) | 2
Paroxysmal atrial fibrillation (Cardiac disorders) | 2
Malaise (General disorders) | 2
Neutrophil count decreased (Investigations) | 7
Creatinine increased (Investigations) | 4
Upper Respiratory infection (Infections and infestations) | 5
Aspartate aminotransferase increased (Investigations) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Headache (Nervous system disorders) | 4
White blood cell decreased (Investigations) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Dizziness (Nervous system disorders) | 3
Sinusitis (Infections and infestations) | 2
Stomach pain (Gastrointestinal disorders) | 3
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
Intermittent hemorhoidal hemorrhage (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 6
Allergic reaction (Immune system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Edema Face (General disorders) | 1
Localized edema (General disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Aortic valve disease (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT01125176/Prot_SAP_000.pdf